CLINICAL TRIAL: NCT00125801
Title: Breakthrough Cancer Pain: A Randomized Trial Comparing Oral Morphine Immediate Release and Self-Administration of Subcutaneous Hydromorphone Using an Injection Pen
Brief Title: The Pain Pen for Breakthrough Cancer Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Dr. Joost L.M. Jongen, Erasmus MC
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMC 02-115
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Neoplasms; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Subcutaneous hydromorphone delivered by pain pen — Subcutaneous hydromorphone delivered by pain pen during breakthrough pain episodes, at max 4 daily. Dose established by opioid conversion from baseline opioids.

SUMMARY:
The purpose of this study is to see whether injection of hydromorphone through a subcutaneous injection device is more effective in treating breakthrough cancer pain than oral morphine.

DETAILED DESCRIPTION:
Breakthrough pain is an exacerbation of severe pain that occurs on a background of otherwise controlled pain. Breakthrough pain is common in patients with advanced cancer. Current medications to treat breakthrough pain include oral immediate release opioid formulations and more recently oral transmucosal fentanyl citrate.

The pain pen study is a randomized controlled double blind cross-over study comparing the efficacy of oral immediate release morphine with that of subcutaneous hydromorphone, injected through a so called pain pen, on breakthrough pain in cancer patients. Preliminary experience with the pain pen suggests that it has a more rapid time of onset of pain relief than oral formulations.

ELIGIBILITY:
Inclusion Criteria:

* Stable cancer pain requiring the equivalent of 60-1000 mg oral morphine/day
* 1-4 breakthrough pain episodes/day
* Patients must be able, in the opinion of the investigator, to fully comply with trial requirements
* Patients who have given written informed consent

Exclusion Criteria:

* Uncontrolled pain
* Women who are pregnant, lactating or intend to become pregnant
* Cardiopulmonary disease that would increase the risk of opioids
* Neurologic or psychiatric disease that would compromise data collection
* Recently started chemotherapy or radiotherapy in as far as it would be effective in lowering breakthrough pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference (PID) at t=15 minutes | t=15 minutes

SECONDARY OUTCOMES:
PID 5' | 5 min
PID 30' | 30 min
PID 45' | 45 min
PID 60' | 60 minutes
time to onset of meaningful pain relief | time to onset
global efficacy rating at 60' | 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Joost L. Jongen, MD, Principal Investigator — Dept. Neurology, Erasmus MC
Locations (1):
- Dept. Neurology, Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Background] Enting RH, Mucchiano C, Oldenmenger WH, Fritzon M, Wallen A, Goslinga-van der Gaag S, Sillevis Smitt PA, Delhaas E. The "pain pen" for breakthrough cancer pain: a promising treatment. J Pain Symptom Manage. 2005 Feb;29(2):213-7. doi: 10.1016/j.jpainsymman.2004.05.010. PMID 15733812
- See also: Related Info — http://www.erasmusmc.nl/neurologie/